CLINICAL TRIAL: NCT00159497
Title: Bone Remodeling Around HA-coated Acetabular Cups.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ON-04-001-MBL
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-03

CONDITIONS: Coxarthrosis
Keywords: THA
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard porouscoated Trilogy Cup
  Interventions: Device: porous coated Trilogy®
- 2 (Experimental): HA coated Trilogy cup
  Interventions: Device: Trilogy Calcicoat®

INTERVENTIONS:
Device: porous coated Trilogy® — THA
  Other Names: Zimmer
  Arms: 1
Device: Trilogy Calcicoat® — THA
  Other Names: Zimmer
  Arms: 2

SUMMARY:
This study was designed to investigate the influence of HA-coating on bone remodeling around the cup in cementless THA.

100 patients gave informed consent to participate in a controlled randomized study between porous coated Trilogy® versus Trilogy Calcicoat®. The cup was inserted in press-fit fixation. The femoral component was a cementless porous coated titanium alloy stem (Bi-Metric®), with a modular 28 mm CrCo head. Effect parameters were Harris Hip Score (HHS) and Bone Mineral Density (BMD) determined by DEXA scanning.

Measurements revealed no difference between the two groups after 3 years, neither in clinical outcome nor in terms of periprosthetic bone density. Patients with Body Mass Index above normal regained more bone mineral than patients with normal weight. This finding supports the assumption that load is beneficial to bone remodeling. Advantages of better sealing of the bone-prosthesis interface, preventing polyethylene induced osteolysis, may still be anticipated for the 7 or 12 year follow-up examinations

DETAILED DESCRIPTION:
This study was designed to investigate the influence of HA-coating on bone remodeling around the cup in cementless THA.

100 patients gave informed consent to participate in a controlled randomized study between porous coated Trilogy® versus Trilogy Calcicoat®. The cup was inserted in press-fit fixation. The femoral component was a cementless porous coated titanium alloy stem (Bi-Metric®), with a modular 28 mm CrCo head. Effect parameters were Harris Hip Score (HHS) and Bone Mineral Density (BMD) determined by DEXA scanning.

Measurements revealed no difference between the two groups after 3 years, neither in clinical outcome nor in terms of periprosthetic bone density. Patients with Body Mass Index above normal regained more bone mineral than patients with normal weight. This finding supports the assumption that load is beneficial to bone remodeling. Advantages of better sealing of the bone-prosthesis interface, preventing polyethylene induced osteolysis, may still be anticipated for the 7 or 12 year follow-up examinations

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for cementless THA

Exclusion Criteria:

* Medical conditions interfering with bone metabolism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 1998-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes in bone mineral density around the hip prosthesis, measured by DEXA scanning | 8-12 years

SECONDARY OUTCOMES:
Changes in hip performance, measured by Harris Hip Score | 8-12 years

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Laursen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Farsoe, Aalborg University Hospital, Farsø, Northern Jutland, Denmark

REFERENCES:
- See also: The final paper from this trial. — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Retrieve&db=pubmed&dopt=Citation&list_uids=16761153